CLINICAL TRIAL: NCT04671173
Title: Real-Time Muscle Pressure Measurements in Patients at Risk for Acute Compartment Syndrome: A Prospective Cohort Study With Historical Control
Brief Title: Real-Time Muscle Pressure Measurements in Patients at Risk for Acute Compartment Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Hennepin Healthcare Research Institute (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Mitchell Bernstein, Assistant Professor, Departments of Surgery & Pediatric Surgery, McGill University and Head, Pediatric 0Orthopaedic Trauma, Montreal Children's Hospital Orthopaedic Trauma & Limb Deformity Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-6655
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Acute Compartment Syndrome
Keywords: Acute compartment syndrome, minimally invasive, sensor, intracompartmental muscle pressure

STUDY DESIGN:
Intervention Model Description: multi-center, non-randomized, historically controlled, prospective pilot trial of the MY01 device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental arm (only one arm) (Experimental): Only one arm, the participants will all received the device to measure Intra-compartmental pressure after consenting to study participation.
  Interventions: Device: Measurement of the Intra-Compartmental Pressure with the MY01 device

INTERVENTIONS:
Device: Measurement of the Intra-Compartmental Pressure with the MY01 device — All Participants will be monitored for clinical signs of symptoms of ACS, including the 7 Ps at a minimum of every 4-6 hours.
  The Intra-Compartmental Pressure of the anterior compartment of the leg will be monitored with the MY01 device. The device should be inserted five centimeters (5 cm) from the fracture, if possible, in the muscle belly. The affected limb will then be splinted in a standard U-slab with no pressure on the monitored device.

SUMMARY:
The purpose of this trial is to conduct a pilot study that will aid in the design of an evaluation of the clinical benefit of MY01, an FDA cleared device, that allows continuous monitoring of intracompartmental muscle pressure in patients at risk for developing acute compartment syndrome. MY01 has previously been successfully tested on animal and Human cadaver Acute Compartment Syndrome models within the RI MUHC through Department of Defense research Grant (Combat Casualty Care Research Program (CCCRP). This trial is supported by the same grant, as the next phase of the overall project.

This is a multi-center, non-randomized, historically controlled, prospective trial of the MY01 device. A cohort of 50 participants will be prospectively enrolled with two weeks follow up to document clinical benefit of the device. Results from this study will be used to inform the design of a larger study designed to demonstrate the clinical benefit of the MY01 device in the early diagnosis of ACS.

The role of each organisation within the trial are detailed below:

* Research Institute of McGill University Health Centre (RI MUHC): study coordination and data analysis (no recruitment activity will take place in the MUHC).
* Hennepin Healthcare: participants recruitment
* Vanderbilt University Medical Centre: participants recruitment

DETAILED DESCRIPTION:
Research Plan

The purpose of this trial is to conduct a pilot study that will inform the design of a trial to evaluate the clinical benefit of MY01, a FDA cleared device that allows continuous monitoring of intracompartmental muscle pressure in patients at risk for developing acute compartment syndrome. The MY01 device is a digitally connected device with a companion mobile app designed to continuously monitor intracompartmental pressure, outputting the results to the mobile app, where clinicians can track the pressure in real time.

There are several goals of this study. Fifty patients with high-energy injuries to the proximal leg and tibial shaft will be prospectively studied and compared to a cohort of historical controls. We want to evaluate the feasibility of collecting data related to the diagnosis of ACS and the measurement of its associated complications. We will also use this data to attempt to assign a modified Boyers grade to a cohort of prospectively enrolled patients and historical controls. Clinical validation of the modified Boyers grade will represent a large step forward in compartment syndrome research, since it will bring an objective assessment of severity to the diagnosis of acute compartment syndrome.

These control patients are to be obtained from several cohorts of patients:

1- Data collected for 3 Retrospective studies on tibial fractures and dislocations resulting in acute compartment syndrome completed in Montreal General Hospital, Vanderbilt University Health Centre and Hennepin Healthcare. The data received from those existing studies will be de-identified.

2 - Patients treated in the PACS study previously funded by DOD and run by METRC.

3- Trauma Quality Programs Participant Use File (TQP) data.

Another goal is to assess the reoperation rates, for limb salvage or amputation among patients that undergo continuous monitoring of ICP using the MY01 monitor relative to a cohort of historical controls who did not receive continuous monitoring.

Primary Research Outcome

Assess the reoperation rate and number of operative procedures for all surgically managed acute compartment syndrome patients.

Secondary Research Outcomes

There are numerous outcomes that are related to the severity of ACS when it is diagnosed. This study will also assess our ability to identify the following secondary outcomes among a cohort of prospectively enrolled patients relative to a cohort of historical controls.

1. Comparison of grades of ACS to the historic controls.
2. Increased proportion of lower ACS outcome grades (Grades 1,2 as per grade)
3. Reduction in time to diagnosis of ACS
4. Improved short-term visual analog pain scores (VAS) for pain in affected limb
5. Reduction in inpatient days
6. Reduction in Skin Grafts
7. Reduction in Major Myectomy
8. Reduction in Anesthesia Time for patients undergoing fasciotomy
9. Clinical ease with which the new compartment pressure monitor was inserted into a muscle compartment, per satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Direct admission to hospital from scene of injury, or if transferred, admitted no more than 12 hours from injury
* High-energy fracture of the tibial plateau (bicondylar or medial fracture - dislocation)
* High energy displaced tibial diaphysis (highly comminuted or segmental fracture, or proximal third of tibia (e.g. GSW to the proximal fibula)) that is felt by the surgeon to have a likelihood of elevated ICP and risk of ACS.

Exclusion Criteria:

1. Frankly contaminated or infected wounds or fractures.
2. Clinical suspicion of acute compartment syndrome requiring urgent fasciotomy at time of presentation to study center.
3. Monitoring could not be initiated within 12 hours of presentation
4. Acute or pre-existing neuropathy in the study limb.
5. Patient is pregnant
6. Patient is a prisoner/incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Reoperation rate (number of re-operation) | 6 weeks
  Assess the reoperation rate for all surgically managed acute compartment syndrome patients following the original fasciotomy.
Number of operative procedures | 6 weeks
  Number of operative procedures for all surgically managed acute compartment syndrome patients.

SECONDARY OUTCOMES:
Comparison of grades of ACS to the historic controls. | 6 weeks
  Comparison of grades of ACS to the historic controls.
Changed proportion of lower ACS outcome grades | 6 weeks
  changed proportion of lower ACS outcome grades (Grades 1,2 as per grade)
Change in time to diagnosis of ACS | 6 weeks
Change in short-term visual analog pain scores (VAS) for pain in affected limb | 6 weeks
Change in inpatient days | 6 weeks
Change in Skin Grafts number | 6 weeks
change in Major Myectomy number | 6 weeks
change in Anesthesia Time for patients undergoing fasciotomy | 6 weeks
Clinician satisfaction survey (percentage) | 6 weeks
  Clinical ease with which the new compartment pressure monitor was inserted into a muscle compartment, per satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Bernstein, Dr, Principal Investigator — Research Institute of McGill University Health Centre (RI MUHC)
Locations (2):
- United States (2):
  - Hennepin County Medical Center - Orthopaedic Research, Minneapolis, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared to other researchers

REFERENCES:
- [Background] Via AG, Oliva F, Spoliti M, Maffulli N. Acute compartment syndrome. Muscles Ligaments Tendons J. 2015 Mar 27;5(1):18-22. eCollection 2015 Jan-Mar. PMID 25878982
- [Background] Shadgan B, Menon M, Sanders D, Berry G, Martin C Jr, Duffy P, Stephen D, O'Brien PJ. Current thinking about acute compartment syndrome of the lower extremity. Can J Surg. 2010 Oct;53(5):329-34. PMID 20858378
- [Background] McQueen MM, Gaston P, Court-Brown CM. Acute compartment syndrome. Who is at risk? J Bone Joint Surg Br. 2000 Mar;82(2):200-3. PMID 10755426
- [Background] Collinge CA, Attum B, Lebus GF, Tornetta P 3rd, Obremskey W, Ahn J, Mirick G, Schmidt A, Spitler C, Coles C, Krause P; Orthopaedic Trauma Association's Evidence-based Quality and Value Committee. Acute Compartment Syndrome: An Expert Survey of Orthopaedic Trauma Association Members. J Orthop Trauma. 2018 May;32(5):e181-e184. doi: 10.1097/BOT.0000000000001128. PMID 29432322
- [Background] Schmidt AH, Bosse MJ, Frey KP, O'Toole RV, Stinner DJ, Scharfstein DO, Zipunnikov V, MacKenzie EJ; METRC. Predicting Acute Compartment Syndrome (PACS): The Role of Continuous Monitoring. J Orthop Trauma. 2017 Apr;31 Suppl 1:S40-S47. doi: 10.1097/BOT.0000000000000796. PMID 28323801
- [Background] Shadgan B, Pereira G, Menon M, Jafari S, Darlene Reid W, O'Brien PJ. Risk factors for acute compartment syndrome of the leg associated with tibial diaphyseal fractures in adults. J Orthop Traumatol. 2015 Sep;16(3):185-92. doi: 10.1007/s10195-014-0330-y. Epub 2014 Dec 28. PMID 25543232
- [Background] McQueen MM, Court-Brown CM. Compartment monitoring in tibial fractures. The pressure threshold for decompression. J Bone Joint Surg Br. 1996 Jan;78(1):99-104. PMID 8898137